CLINICAL TRIAL: NCT00783068
Title: The Effect of the Alpha-7 Nicotinic AChR Agonist GTS-21 on Inflammation and End-organ Dysfunction During Human Endotoxemia
Brief Title: Anti-inflammatory Effects of GTS-21 After LPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: CoMentis (Industry)
Responsible Party: Prof. Dr. J.G. van der Hoeven, Radboud University Nijmegen Medial Centre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL 20388.091.07
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2008-10

CONDITIONS: Endotoxemia; Sepsis; Vagal Activity
Keywords: Endotoxin; GTS-21; Vagal activity; Autonomic balance
MeSH Terms: conditions — Endotoxemia; Sepsis | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTS-21 (Active Comparator): Subjects will be randomized to oral pre-treatment with GTS-21 (150 mg tid 3 days before LPS injection and an oral dose of 150 mg GTS-21 on the morning of the day of the experiment (07:00 AM). Subjects will then receive an oral dose of 150 mg GTS-21 or placebo at 08:00 AM and another oral dose of 150 mg GTS-21 or placebo at 1 hour before LPS administration (t=0).
  Interventions: Drug: GTS-21, [3-(2,4-dimethoxybenzylidene)-anabaseine dihydrochloride]; Drug: Lipopolysaccharide E. Coli 113:H 10:K negative
- Placebo (Placebo Comparator): Subjects will receive placebo 3 day before injection of LPS (150 mg tid) and a single oral dose of 150 mg of placebo the morning of LPS injection (07:00 AM). Subjects will then receive an oral dose of 150 mg placebo at 08:00 AM and another oral dose of 150 mg placebo at 1 hour before LPS administration (t=0).
  Interventions: Drug: Placebo; Drug: Lipopolysaccharide E. Coli 113:H 10:K negative

INTERVENTIONS:
Drug: GTS-21, [3-(2,4-dimethoxybenzylidene)-anabaseine dihydrochloride] — Subjects will receive GTS-21 or placebo 3 day before injection of LPS (150 mg tid) and a single oral dose of 150 mg of GTS-21 or placebo the morning of LPS injection (07:00 AM). Subjects will then receive an oral dose of 150 mg GTS-21 or placebo at 08:00 AM and another oral dose of 150 mg GTS-21 or placebo at 1 hour before LPS administration (t=0)
  Other Names: GTS-21
  Arms: GTS-21
Drug: Placebo — Subjects will receive placebo 3 day before injection of LPS (150 mg tid) and a single oral dose of 150 mg of placebo the morning of LPS injection (07:00 AM). Subjects will then receive an oral dose of 150 mg placebo at 08:00 AM and another oral dose of 150 mg placebo at 1 hour before LPS administration (t=0).
  Other Names: Test
  Arms: Placebo
Drug: Lipopolysaccharide E. Coli 113:H 10:K negative — Subjects will be randomized to oral pre-treatment with GTS-21 (150 mg tid 3 days before LPS injection and an oral dose of 150 mg GTS-21 on the morning of the day of the experiment (07:00 AM). Subjects will then receive an oral dose of 150 mg GTS-21 or placebo at 08:00 AM and another oral dose of 150 mg GTS-21 or placebo at 1 hour before LPS administration (t=0). One hour after ingestion of the last dosage of the study drug, purified LPS prepared from E coli O:113 (2 ng/kg iv) will be injected intravenously.
  Other Names: Endotoxin

SUMMARY:
Rationale: The vagus nerve exerts an anti-inflammatory effect in in vitro and animal experiments. This 'vagal anti-inflammatory pathway' is mediated by the nicotinergic α7nACh receptor that can be selectively stimulated by GTS-21. Activation of the cholinergic anti-inflammatory pathway via vagus nerve stimulation or α7nAChR agonists improves outcome in animal models of endotoxemia, sepsis and experimental arthritis. Up to now, the anti-inflammatory effects of oral administration of GTS-21 in humans in vivo has not been investigated.

Objective: Primary aim: to investigate the anti-inflammatory effects of oral administration of GTS-21 on the inflammatory response in the human endotoxemia model and the subsequent inflammation-induced subclinical organ dysfunction. Secondary aim: to measure the effect of LPS administration in the absence or presence of GTS-21 in human volunteers on vagal nerve activity measured by heart rate variability analysis.

Study design: Double-blind placebo-controlled randomized cross-over intervention study in healthy human volunteers during experimental endotoxemia.

Study population: Non-smoking healthy male volunteers, age 18-35 yrs Intervention: Subjects will be tested in a cross-over design in 2 separate sequential sessions, 2-4 weeks apart. A total of 12 subjects will be randomly assigned to one of two dosing groups in a 1:1 ratio: GTS-21 followed by Placebo n=6, Placebo followed by GTS-21 n=6. Subjects will receive 150mg GTS-21 or placebo orally tid 3 days before LPS injection and an oral dose of 150 mg GTS-21 or placebo the morning of the day of LPS administration (07:00 AM). Subjects will then receive an oral dose of 150 mg GTS-21 or placebo at 08:00 AM and another oral dose of 150 mg GTS-21 or placebo at 1 hour before LPS administration (t=0). Before LPS injection, prehydration will be performed by infusion of 1.5 L 2.5% glucose/0.45% saline solution in 1 hour. One hour after the last dose of GTS-21 or placebo, LPS derived from E coli O:113 will be injected (2 ng/kg iv in 1 minute). There will be a 14 day washout period for patients in all groups. The last group of subjects will be subjected to an identical dose of LPS and placebo at two different moments 2-4 weeks apart to obtain time controls.

Main study parameters/endpoints: Main study endpoint is the concentration of circulating cytokines after LPS in the absence and presence of GTS-21.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: A medical interview and physical examination is part of this study. Approximately 350 ml blood will be withdrawn and urine will be collected. There will be mild discomfort associated with participation in this study, as LPS induces flu-like symptoms for approximately 4 hrs. GTS-21 was found to be well tolerated at a dose of 150 mg three times daily (450 mg/day).

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE: The innate immune response is the first line of defense against invading pathogens(1). This tightly regulated system consists of a wide variety of chemokines, cytokines, cell associated receptors and other mediators orchestrating the initial response to infection. Experimental evidence in the past several years has demonstrated that activation of the efferent vagus nerve has an inhibitory effect on the innate immune response (the cholinergic anti-inflammatory pathway, reviewed in (2,3,4)). The anti-inflammatory effect of the vagal nerve is mediated by the α7 nicotinic acetylcholine receptor (α7nAChR) expressed on macrophages and other cytokine-producing cells (9). Activation of the cholinergic anti-inflammatory pathway with vagus nerve stimulation or α7nAChR agonists improves outcome in animal models of endotoxemia, sepsis and experimental arthritis. This cholinergic anti-inflammatory pathway is the efferent arm of a reflex mechanism that is activated by inflammatory mediators in peripheral tissues signaling through the afferent vagus nerve. Thus, the vagus nerve can relay inflammation signals to the central nervous system and activate an opposing efferent response to inhibit excessive inflammation.

GTS-21 (E-3-(2,4)-dimethoxybenzylidene anabaseine) is a highly specific α7nAchR agonist, that has been developed for the treatment of Alzheimer's disease that has been studied in a few inflammation-related models. In a murine pancreatitis model pre-treatment of the animals with GTS-21 decreased pancreatitis severity and was associated with reduced IL-6 levels and decreased pancreatic neutrophil accumulation (11). Pre-treatment of mice with GTS-21 attenuated systemic TNF concentrations after injection with LPS and increases survival (12,13). Similarly, GTS-21 inhibited blood levels of the inflammatory mediator High Mobility Group Box 1 (HMGB1) and improved survival of mice after cecal ligation and puncture.(13). Recently, we have shown that stimulation of the α7nAChR by the highly selective agonist GTS-21 leads to a dramatic dose-dependent inhibition of pro-inflammatory cytokine release induced by stimulation of various Toll-like receptors (TLR) in human whole blood (Kox et al, submitted). This inhibitory effect of GTS-21 was not specific for the TLR-agonist used and GTS-21 inhibited pro-inflammatory cytokine production stronger than nicotine at equimolar concentrations. Moreover, the production of the anti-inflammatory cytokine IL-10 was not inhibited, but even significantly stimulated. Therefore, stimulation of the α7nAChR by GTS-21 results in a profound anti-inflammatory shift of the pro-/anti-inflammatory balance. So far, no data are available on the anti-inflammatory effects of GTS-21 in humans in vivo.

The human endotoxemia model is widely used to study inflammation in humans in vivo. Systemic inflammation is induced by low-dose infusion of Escherichia coli lipopolysaccharide (LPS) in healthy volunteers, resulting in flu-like symptoms, increased production of C-reactive protein and increased concentrations of pro- and anti-inflammatory cytokines. The "human endotoxemia model" permits elucidation of key players in this proinflammatory response in humans in vivo and it serves as a useful tool to investigate potential novel therapeutic strategies in a standardized setting.

GTS-21 was developed as a novel agent in the treatment of Alzheimer's disease. Until date, 87 healthy male volunteers were enrolled in four Phase I studies that assessed the safety, tolerability, pharmacokinetics, and effects on cognitive function of oral administration of GTS-21 of which 77 subjects received GTS-21 and 10 subjects received placebo. GTS-21 was found to be well tolerated up to a dose of 150 mg three times daily (450 mg/day) in healthy male subjects. The most common adverse event was headache, which occurred in 27% of subjects in the GTS-21 group compared to 21% of subjects in the placebo group. There were no serious adverse events, or severe adverse events reported during these studies. In one patient in the GTS-21 group transient mild elevation of liver enzymes was detected, without signs of hepatic dysfunction.

PRIMARY AIM: Primary aim of the present study is to investigate the putative anti-inflammatory effects of oral administration of GTS-21 on the inflammatory response and subsequent subclinical organ dysfunction in the human endotoxemia model. Secondary aim is to measure the effect of LPS administration in the absence and presence of GTS-21 in human volunteers on vagal nerve activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 35 yrs
* Male
* Healthy

Exclusion Criteria:

* Use of any medication
* Smoking
* History, signs or symptoms of cardiovascular disease
* (Family) history of cerebrovascular disease
* Previous vagal collapse
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinin >120 μmol/l)
* Liver enzyme abnormalities or positive hepatitis serology
* Positive HIV test

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To investigate the putative anti-inflammatory effects of oral administration of GTS-21 on the inflammatory response and subsequent subclinical organ dysfunction in the human endotoxemia model. | 24 hours after LPS

SECONDARY OUTCOMES:
To measure the effect of LPS administration in the absence and presence of GTS-21 in human volunteers on vagal nerve activity. | 24 hours afte LPS
Concentration of pro- and anti-inflammatory cytokines. | 24 hours after LPS
AChR and TLR expression on circulating monocytes | 24 ours after LPS
Concentration of HMGB-1 | 24 hours after LPS
Leucocyte number, C-reactive protein concentrations | 24 hours after LPS
Hemodynamic parameters, Severity of clinical symptoms | 24 hours after LPS
Markers of endothelial damage (adhesion molecules) | 24 hours after LPS
Urine excretion of markers of proximal (GSTA1-1) and distal (GSTP1-1) renal tubular damage | 24 hours after LPS
Vagal activity as measured by heart rate variability analysis | 24 hours after LPS
Body temperature | 24 hours after LPS
Additional blood samples will be drawn for measurement of: TLR-expression, Genetics; micro array analyses and determination of intercellular signalling pathways. | 24 hours after LPS

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands